CLINICAL TRIAL: NCT05675384
Title: SAFETY AND EFFECTIVENESS OF TRANSCUTANEOUS ELECTRICAL NERVE STIMULATION (TENS)-ASSISTED WEIGHT MANAGEMENT (THE ELIRA SYSTEM) AS COMPARED TO A SHAM DEVICE
Brief Title: Safety & Effectiveness of TENS Weight Management Compared to a Sham
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Elira, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CD-006
Record Dates: First submitted 2022-12-29; First posted 2023-01-09 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2022-12

CONDITIONS: Obesity, Mild
MeSH Terms: conditions — Obesity; Lymphoma, Follicular

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- TENS Active Treatment (Experimental): Transcutaneous Electrical Nerve Stimulation (TENS)-Assisted Weight Management (The Elira System)
  Interventions: Device: TENS Active Treatment
- Sham Control Device (Sham Comparator): Sham TENS unit that provides no actual therapy
  Interventions: Device: Sham Device

INTERVENTIONS:
Device: TENS Active Treatment — Using a 7-day/week wearable TENS device controlled by a Smart Phone App combined with moderate intensity lifestyle therapy,
  Arms: TENS Active Treatment
Device: Sham Device — Using the sham (control) device combined with a moderate intensity lifestyle follow-up
  Arms: Sham Control Device

SUMMARY:
This is a multicenter, randomized, blinded, parallel group, controlled study intended to evaluate the safety and effectiveness of treating overweight and Class 1 obese patients with the Elira System (TENS active treatment) combined with a moderate intensity lifestyle follow-up compared to participants using the sham (control) device combined with a moderate intensity lifestyle follow-up

DETAILED DESCRIPTION:
This is a multicenter, randomized, blinded, parallel group, controlled study intended to evaluate the safety and effectiveness of treating overweight and Class 1 obese patients with the Elira System (TENS active treatment) combined with a moderate intensity lifestyle follow-up compared to participants using the sham (control) device combined with a moderate intensity lifestyle follow-up. The objective is to demonstrate the effectiveness of the Elira System combined with a moderate intensity lifestyle therapy program compared to a sham device combined with a moderate intensity lifestyle therapy program control group at 3-months on weight management for participants who are overweight and/or with Class 1 obesity.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is between 18 - 65 years of age inclusive.
2. Participant has a BMI of 25 to < 35 kg/ m2.
3. Participant has signed the informed consent form and is able to comply with study protocol and adhere to study visit schedule.
4. Participant is able to use a touch screen handheld smart phone.
5. Participant has Wi-Fi internet access for the duration of the study.
6. Participant is fluent in English or Spanish and can complete questionnaires.
7. Females of childbearing potential (FOCBP) must have a negative urine pregnancy test at screening and enrollment visit and agree to using birth control to avoid pregnancy during the trial, prior to placement of assigned treatment device.
8. Participant agrees to adhere to diet & exercise recommendations throughout study duration.
9. Participant is willing and able to adhere to assigned therapy throughout the study duration.
10. Participant has not participated in any clinical trial (except a registry) within the last 30 days.-

Exclusion Criteria:

1. Participant has any known gastrointestinal disorder that in the opinion of the Investigator precludes enrollment into the trial.
2. Participant has had a prior bariatric surgical procedure, endoscopic bariatric therapy, or surgery on the stomach.
3. Participant has any significant multisystem disease in the opinion of the Investigator.
4. Participant is a Type 2 diabetic.
5. Participant has a history of significant cardiac arrhythmia, ectopy, or significant cardiovascular disease.
6. Participant has an existing implanted electrical stimulator (e.g., pacemaker, AICD, cochlear implant).
7. For female participants: planned pregnancy within 6 months from study start, active pregnancy, or currently breast feeding.
8. Participant has current and/or a history of cancer with the exception of non-melanoma skin cancer or cervical carcinoma in situ < 3 years before study enrollment.
9. Participant has had a weight change of ± 5% of his/her Total Body Weight in the 3 months prior to screening.
10. Participant has an uncontrolled psychiatric disorder.
11. Participant has a diagnosed neurological disease.
12. Participant has a skin disorder affecting the thoracic dermatomes.
13. Participant has active/has ever had shingles in the abdominal area.
14. Participant has abdominal surgery or other scars which may interfere with TENS stimulation in the opinion of the PI.
15. Participant has known allergic reaction to materials in the TENS electrodes and/or is otherwise unable to tolerate stimulation with the wearable TENS system. This includes known allergies or sensitivity to latex, nickel and/or hydrogels.
16. Participant has a history of sensitive skin, including eczema wheel-and-flare or other skin irritation, per PI discretion.
17. Participant is actively participating or unwilling to discontinue participation in another weight loss program. (Participants may not enroll in paid or unpaid programs that involve inperson or online coaching during the course of the Elira study.)
18. Participant has a history of eating disorders (Bulimia, Binge Eating, Night Eating Syndrome, Compulsive Overeating) and/or screens positive for Binge Eating as measured by the Binge Eating Score (BES) Questionnaire.
19. Participant has taken weight loss medications including but not limited to OTC medications or any other medication known to cause weight loss or weight gain within the 2 months prior to enrollment.
20. Participant is planning any major medical treatments or surgeries that could cause weight loss during the study.
21. Participant works night shift or rotating night shifts that impact scheduled daylight mealtimes.
22. Inability to walk at least 0.8 kilometers per day (10 minutes of continuous walking).
23. Current smoker or user of nicotine product or smoking cessation within 1 year of the screening date.
24. History of treatment for or current abuse of drugs or alcohol.
25. A score of 10 or higher on the Patient Health Questionnaire 9 (PHQ-9), demonstrating moderate depression.
26. Any participant that the Investigator considers inappropriate for the study for medical reasons.
27. Participant is taking Topiramate, Adderall, or Ritalin within the 6 months prior to enrollment.
28. Participant is on drug therapy which may alter antral motility or appetite, per Investigator discretion within the 2 months prior to enrollment.
29. History of cirrhosis or pancreatitis.
30. History of COPD or other pulmonary disease that restricts exercise tolerance.
31. Immunocompromised due to medications or disease or HIV positive.
32. History of severe Covid-19 symptoms requiring hospitalization or history of Covid-19 infection with unresolved symptoms.
33. TSH levels > 10mU/L or < 0.1 mU/L.
34. Prior participation in an Elira sponsored study.
35. A current member of the participant's household has been randomized into the Elira 3 study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 395 (Actual)
Dates: Start 2022-07-29 (Actual); Primary Completion 2024-07-23 (Actual); Study Completion 2024-07-23 (Actual)

PRIMARY OUTCOMES:
A difference in Percent Total Body Weight Loss (%TBWL) | Three Months
  A difference in Percent Total Body Weight Loss (%TBWL) of greater than 0 (true mean percent of 2%) at 3-months in the Elira System (active) treatment group when compared to the sham (control) group who complete 3-months of treatment
A responder rate of at least 35% in the active treatment | Three Months
  A responder rate of at least 35% in the active treatment participants who complete 3-months of treatment, calculated as the percentage achieving at least a 5% TBWL at 3-months

SECONDARY OUTCOMES:
Changes in appetite as measured by Appetite Visual Analogue Scale (VAS) | Three Months
  Changes in appetite as measured by Appetite Visual Analogue Scale (VAS) from Baseline to 3-months in the active treatment group compared to the sham control group
Changes in BMI | Three Months
  Changes in BMI from Baseline to 3-months in the active treatment group compared to the sham control group
Changes in eating behaviors as measured by TFEQ scores | Three Months
  Changes in eating behaviors as measured by TFEQ scores from Baseline to 3-months in the active treatment group compared to the sham control group
Impact of weight on quality of life (IWQOL-Lite) scores | Three Months
  Impact of weight on quality of life (IWQOL-Lite) scores from Baseline to 3-months in in the active treatment group compared to the sham control group

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Honor Health, Scottsdale, Arizona
  - EmVenio, Santa Monica, California
  - A New You, Miami, Florida
  - Advanced Research for Health Improvement, LLC (ARHI), Naples, Florida
  - Washington University, St Louis, Missouri
  - West County OB/GYN Specialists, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: No